CLINICAL TRIAL: NCT04972552
Title: Watermelon/UBIQuinone Study (WUBI-Q Trial)
Brief Title: Watermelon/UBIQuinone Study
Acronym: WUBI-Q
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 21-34366
Record Dates: First submitted 2021-07-02; First posted 2021-07-22 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: 2x2 placebo-controlled factorial trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed by a pharmacy and investigators will not know the assignment until trial completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Watermelon Diet & Coenzyme Q10 (Active Comparator): 800-1200 mg of coenzyme Q10 daily plus diet high in watermelon
  Interventions: Dietary Supplement: coenzyme Q10; Other: Watermelon diet
- Usual Diet & Coenzyme Q10 (Active Comparator): 800-1200 mg of coenzyme Q10 daily plus no watermelon in diet
  Interventions: Dietary Supplement: coenzyme Q10; Other: Usual Diet
- Watermelon Diet & Placebo (Placebo Comparator): Placebo pill plus diet high in watermelon
  Interventions: Other: Watermelon diet; Other: Placebo
- Usual Diet & Placebo (Placebo Comparator): Placebo pill plus no watermelon in diet
  Interventions: Other: Usual Diet; Other: Placebo

INTERVENTIONS:
Dietary Supplement: coenzyme Q10 — Participants will take 800-1200 mg of coenzyme Q10 capsule per day
  Other Names: CoQ10
  Arms: Usual Diet & Coenzyme Q10; Watermelon Diet & Coenzyme Q10
Other: Watermelon diet — Participants will be asked to eat watermelon at a minimum of one meal per day 3-5 days a week
  Arms: Watermelon Diet & Coenzyme Q10; Watermelon Diet & Placebo
Other: Usual Diet — Participants will be asked to eat a usual diet but not eat any watermelon as part of their usual diet
  Arms: Usual Diet & Coenzyme Q10; Usual Diet & Placebo
Other: Placebo — Participants will be asked to take 800-1200 mg of a placebo capsule per day
  Arms: Usual Diet & Placebo; Watermelon Diet & Placebo

SUMMARY:
The objective of the proposed pilot trial is to determine the feasibility and safety of increasing watermelon consumption, with or without coenzyme Q supplementation in patients after kidney transplantation on kidney function and urinary protein excretion.

DETAILED DESCRIPTION:
While many observational studies have examined the effects of consuming watermelon in patients without chronic kidney disease, there have been few studies on the consumption of a diet high in watermelon as a means of improving kidney function or reducing protein in the urine. Coenzyme Q is also recognized as a supplement that has benefits for heart health and has anti-oxidative effects, but whether it could be used to improve kidney function or reduce protein in the urine has not been thoroughly examined, especially in the kidney transplant population. The objective of the proposed pilot trial is to determine the feasibility and safety of increasing watermelon consumption, with or without coenzyme Q supplementation in patients after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Received a kidney transplant in the last four weeks
* History of dialysis dependency prior to kidney transplant
* Able to provide informed consent
* Not currently consuming a high-watermelon diet or taking co-enzyme Q10
* Not underweight (body mass index <19 kg/m2)
* Not enrolled in any other interventional trial
* Planning to return for follow-up at UCSF (or willing to return for study visits)

Exclusion Criteria:

* < 18 years of age at the time of transplant
* Preemptive transplantation
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients who complete the study after randomized assignment | Measured at the 20 weeks mark
  We will determine the number of patients who drop out of the study following randomized assignment
Number of participants who develop adverse safety events (including low systolic blood pressure or hyperkalemia) during participation in the study | Measured from 0-20 weeks
  We will measure the number of patients who develop low blood pressure and high potassium levels (hyperkalemia) following randomized assignment. Low blood pressure will be defined as systolic blood pressure < 90 mmHg; hyperkalemia will be defined as serum potassium > 5.5 meq/L

SECONDARY OUTCOMES:
Mean change in weight from baseline to 20 weeks | Baseline to 20 weeks
  We will check for a change in weight, measured in kg, at the start and end of the intervention period.
Changes in amount of protein excretion in the urine over a 20-week period | Baseline to 20 weeks
  We will check for a change in urine protein/creatinine ratio (g/g) at the start and end of the intervention period.
Proportion of participants with an eGFR < 60 mL/min/1.73 m2 | Baseline to 20 weeks
  We will assess kidney function outcomes at week 20
Amount of interstitial fibrosis and tubular atrophy | At 20 weeks (cross-sectional)
  We will compare the degree of interstitial fibrosis or tubular atrophy (as a percentage on a biopsy specimen) based on kidney biopsy results.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ku, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lum T, Connolly M, Marx A, Beidler J, Hooshmand S, Kern M, Liu C, Hong MY. Effects of Fresh Watermelon Consumption on the Acute Satiety Response and Cardiometabolic Risk Factors in Overweight and Obese Adults. Nutrients. 2019 Mar 12;11(3):595. doi: 10.3390/nu11030595. PMID 30870970
- [Background] Hong MY, Hartig N, Kaufman K, Hooshmand S, Figueroa A, Kern M. Watermelon consumption improves inflammation and antioxidant capacity in rats fed an atherogenic diet. Nutr Res. 2015 Mar;35(3):251-8. doi: 10.1016/j.nutres.2014.12.005. Epub 2015 Jan 3. PMID 25631716
- [Background] Figueroa A, Wong A, Jaime SJ, Gonzales JU. Influence of L-citrulline and watermelon supplementation on vascular function and exercise performance. Curr Opin Clin Nutr Metab Care. 2017 Jan;20(1):92-98. doi: 10.1097/MCO.0000000000000340. PMID 27749691
- [Background] Figueroa A, Sanchez-Gonzalez MA, Wong A, Arjmandi BH. Watermelon extract supplementation reduces ankle blood pressure and carotid augmentation index in obese adults with prehypertension or hypertension. Am J Hypertens. 2012 Jun;25(6):640-3. doi: 10.1038/ajh.2012.20. Epub 2012 Mar 8. PMID 22402472
- [Background] Rivara MB, Yeung CK, Robinson-Cohen C, Phillips BR, Ruzinski J, Rock D, Linke L, Shen DD, Ikizler TA, Himmelfarb J. Effect of Coenzyme Q10 on Biomarkers of Oxidative Stress and Cardiac Function in Hemodialysis Patients: The CoQ10 Biomarker Trial. Am J Kidney Dis. 2017 Mar;69(3):389-399. doi: 10.1053/j.ajkd.2016.08.041. Epub 2016 Dec 4. PMID 27927588
- [Background] Yu JH, Lim SW, Luo K, Cui S, Quan Y, Shin YJ, Lee KE, Kim HL, Ko EJ, Chung BH, Kim JH, Chung SJ, Yang CW. Coenzyme Q10 alleviates tacrolimus-induced mitochondrial dysfunction in kidney. FASEB J. 2019 Nov;33(11):12288-12298. doi: 10.1096/fj.201900386RR. Epub 2019 Aug 20. PMID 31431058
- [Background] Dlugosz A, Kuzniar J, Sawicka E, Marchewka Z, Lembas-Bogaczyk J, Sajewicz W, Boratynska M. Oxidative stress and coenzyme Q10 supplementation in renal transplant recipients. Int Urol Nephrol. 2004;36(2):253-8. doi: 10.1023/b:urol.0000034652.88578.a8. PMID 15368706
- [Background] Yeung CK, Billings FT 4th, Claessens AJ, Roshanravan B, Linke L, Sundell MB, Ahmad S, Shao B, Shen DD, Ikizler TA, Himmelfarb J. Coenzyme Q10 dose-escalation study in hemodialysis patients: safety, tolerability, and effect on oxidative stress. BMC Nephrol. 2015 Nov 3;16:183. doi: 10.1186/s12882-015-0178-2. PMID 26531095
- [Background] Shanely RA, Nieman DC, Perkins-Veazie P, Henson DA, Meaney MP, Knab AM, Cialdell-Kam L. Comparison of Watermelon and Carbohydrate Beverage on Exercise-Induced Alterations in Systemic Inflammation, Immune Dysfunction, and Plasma Antioxidant Capacity. Nutrients. 2016 Aug 22;8(8):518. doi: 10.3390/nu8080518. PMID 27556488